CLINICAL TRIAL: NCT01515345
Title: Individualizing Dual Antiplatelet Therapy After Percutaneous Coronary Intervention - The IDEAL-PCI Registry
Acronym: IDEAL-PCI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Franz Josef Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Guenter Christ, Univ. Prof. Dr., Kaiser Franz Josef Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDEAL-PCI protocol 1.0
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Platelet Inhibition; Coronary Stent Implantation
Keywords: clopidogrel-nonresponder; stent thrombosis
MeSH Terms: interventions — Prasugrel Hydrochloride; Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard therapy (Active Comparator): standard dual antiplatelet therapy after PCI for all patient populations (stable CVD and ACS)
  Interventions: Drug: Clopidogrel
- individualized therapy (Experimental): dual antiplatelet therapy modified according to clopidogrel on-treatment platelet reactivity measured by Multiplate Analyzer
  Interventions: Drug: prasugrel or ticagrelor

INTERVENTIONS:
Drug: prasugrel or ticagrelor — prasugrel 10mg od for 12 month ticagrelor 90mg td for 12 month
  Other Names: Efient; Brilique
  Arms: individualized therapy
Drug: Clopidogrel — clopidogrel 75mg od for 12 month
  Other Names: Plavix
  Arms: standard therapy

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a routine individualized antiplatelet therapy after coronary stent implantation by evaluating "on-treatment" platelet reactivity with Multiple Electrode Aggregometry (MEA, Multiplate® Analyzer).

DETAILED DESCRIPTION:
Depending on the clinical presentation patients are treated according to standard operating procedures in our department. The earliest, 12 hours after an initial clopidogrel-loading dose (600mg)"on-treatment" platelet reactivity will be determined by Multiple Electrode Aggregometry (MEA, Multiplate® Analyzer), a point of care assay. In case of high residual platelet reactivity (i.e. ≥ 50U), patients are switched according to a therapeutic algorithm to either prasugrel (Efient®), or in case of contraindication (i.e. stroke) to ticagrelor (Brilique®), or in case of contraindication (intracranial hemorrhage) reloaded with clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive PCI patients with stent implantation of our institution

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guenter Christ, MD, Principal Investigator — Kaiser Franz Josef Hospital
Locations (1):
- Kaiser Franz Josef Hospital, Vienna, Vienna, Austria

REFERENCES:
- [Background] Sibbing D, Braun S, Morath T, Mehilli J, Vogt W, Schomig A, Kastrati A, von Beckerath N. Platelet reactivity after clopidogrel treatment assessed with point-of-care analysis and early drug-eluting stent thrombosis. J Am Coll Cardiol. 2009 Mar 10;53(10):849-56. doi: 10.1016/j.jacc.2008.11.030. PMID 19264241
- [Background] Bonello L, Camoin-Jau L, Arques S, Boyer C, Panagides D, Wittenberg O, Simeoni MC, Barragan P, Dignat-George F, Paganelli F. Adjusted clopidogrel loading doses according to vasodilator-stimulated phosphoprotein phosphorylation index decrease rate of major adverse cardiovascular events in patients with clopidogrel resistance: a multicenter randomized prospective study. J Am Coll Cardiol. 2008 Apr 8;51(14):1404-11. doi: 10.1016/j.jacc.2007.12.044. PMID 18387444
- [Background] Price MJ, Berger PB, Teirstein PS, Tanguay JF, Angiolillo DJ, Spriggs D, Puri S, Robbins M, Garratt KN, Bertrand OF, Stillabower ME, Aragon JR, Kandzari DE, Stinis CT, Lee MS, Manoukian SV, Cannon CP, Schork NJ, Topol EJ; GRAVITAS Investigators. Standard- vs high-dose clopidogrel based on platelet function testing after percutaneous coronary intervention: the GRAVITAS randomized trial. JAMA. 2011 Mar 16;305(11):1097-105. doi: 10.1001/jama.2011.290. PMID 21406646
- [Derived] Christ G, Siller-Matula JM, Francesconi M, Dechant C, Grohs K, Podczeck-Schweighofer A. Individualising dual antiplatelet therapy after percutaneous coronary intervention: the IDEAL-PCI registry. BMJ Open. 2014 Oct 31;4(10):e005781. doi: 10.1136/bmjopen-2014-005781. PMID 25361837
- See also: Related Info — http://www.multiplate.net

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all consecutive PCI patients with stent implantation or drug eluting balloon dilation in our institution until June 2012
Period: Overall Study
Arm/Group | Standard Therapy | Individualized Therapy
Started | 665 | 343
Completed | 664 | 343
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy | Individualized Therapy | Total
Number analyzed (Participants) | 665 | 343 | 1008
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 333 | 169 | 502
  >=65 years | 332 | 174 | 506
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12) | 64 (12) | 65 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 120 | 303
  Male | 482 | 223 | 705
Region of Enrollment [Number; unit: participants]
  Austria | 665 | 343 | 1008

OUTCOME MEASURES:

1. Primary Outcome: Definite Stent Thrombosis
Description: The angiographic or pathological confirmation of stent thrombosis is called "definite stent thrombosis"
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Standard Therapy | Individualized Therapy
Number analyzed (Participants) | 664 | 343
participants | 1 | 0

2. Primary Outcome: Any Bleeding Event
Description: Bleeding classified by the TIMI hemorrhage classification scheme:
  Minor: any clinically overt sign of hemorrhage (including imaging) that is associated with a hemoglobin drop of 3 to < 5 g/dL
  Major: (1) if it is intracranial, or (2) clinically significant overt signs of hemorrhage associated with a drop inhemoglobin of > 5 g/dL
Time Frame: 30days
Measure: Number; unit: participants
Arm/Group | Standard Therapy | Individualized Therapy
Number analyzed (Participants) | 664 | 343
participants | 17 | 9

3. Secondary Outcome: Probable Stent Thrombosis
Description: Probable stent thrombosis is considered to have occurred in case of
  1. any unexplained death within the first 30 days.
  2. any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause, irrespective of the time after the index procedure
Time Frame: 30days
Measure: Number; unit: participants
Arm/Group | Standard Therapy | Individualized Therapy
Number analyzed (Participants) | 664 | 343
participants | 2 | 0

ADVERSE EVENTS:
Description: it was not intended to collect adverse events, other than SAEs
Arm/Group | Standard Therapy | Individualized Therapy
Serious Adverse Events (participants affected / at risk) | 26/664 | 18/343
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (N=664) | Individualized Therapy (N=343)
Definite stentthrombosis (Cardiac disorders) | 1 (1) | 0 (0)
probable Stentthrombosis (Cardiac disorders) | 2 (2) | 0 (0)
Cardiovascular death (Cardiac disorders) | 6 (6) | 9 (9)
Bleeding (TIMI major) (Cardiac disorders) | 6 (6) | 4 (4)
Bleeding (TIMI minor) (Cardiac disorders) | 11 (11) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No